CLINICAL TRIAL: NCT04046133
Title: Phase 1b/II Trial of Checkpoint Inhibitor (Pembrolizumab an Anti PD-1 Antibody) Plus Standard IMRT in HPV Induced Stage III/IV Carcinoma of Anus
Brief Title: Phase 1b/II Trial of Pembrolizumab Plus IMRT in Stage III/IV Carcinoma of Anus
Acronym: CORINTH
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cardiff University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPON 1529-16
Record Dates: First submitted 2018-01-29; First posted 2019-08-06 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Anal Cancer Stage III A; Anal Cancer Stage III B
MeSH Terms: conditions — Anus Neoplasms | interventions — pembrolizumab; Radiotherapy; Drug Therapy; Mitomycin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- pembrolizumab (Experimental): Patients with locally advanced (stage IIIA/B, T3/T4, any N, M0) anal cancer will receive pembrolizumab, an immune checkpoint inhibitor, concomitantly with standard CRT.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab, an immune checkpoint inhibitor, concomitantly with standard CRT in patients with locally advanced T3/4 anal cancer.
  Other Names: Radiotherapy; Chemotherapy (Mytomycin or Mitomycin and Capecitabine)

SUMMARY:
The CORINTH trial is for patients with more advanced (stage 3 and 4) anal cancer. The numbers of patients with anal cancer is increasing and only 65% patients with this later stage anal cancer have not had a recurrence 3 years after treatment. Anal cancer responds well to chemo-radiation (CRT) and this would be the treatment used for standard clinical care. The chemotherapy in CORINTH will be the same as standard of care (Mitomycin and 5FU or capecitabine) and the radiotherapy (RT) will be delivered using a technique where the dose intensity of RT can be modulated for different areas of the tumor (Intensity Modulated RT - IMRT). Translational samples (tissue blocks and blood) will be collected at baseline with further blood and tissue samples during and after treatment.

Pembrolizumab, a relatively new drug, is a monoclonal antibody that enhances the body's immune response to cancer cells by acting on a receptor on the surface of T-cells called Programmed Death -1 (PD-1). The CORINTH study aims to see whether pembrolizumab, can be added safely to standard CRT. We will explore how safe the combination is and how well tolerated it is for patients with stage 3 and 4 anal cancer. If it is tolerable more patients will be treated to see if there is a similar or better clinical response.

The trial is designed in 3 groups of patients. All patients will receive eight infusions of pembrolizumab at three weekly intervals. Each infusion lasts approximately 1 hour. The first group will not get pembrolizumab until they have already had 4 weeks of CRT (Day 29). As long as this is not found to cause too many extra side effects, the next group will have infusions at the beginning of the third week of CRT. The final group (cohort 3) will start their pembrolizumab with the first day of CRT i.e. Day 1.

Initially each group will have 6 patients. Provided each group of patients finds the treatment tolerable and it is safe, more patients will be recruited into the group that receives the pembrolizumab earliest during their CRT. This will add further credence to the safety and tolerability of the combination and may provide a signal of how effective this treatment might be in improving outcomes for patients with more advanced anal cancer.

DETAILED DESCRIPTION:
CORINTH is a multi center trial with a single arm. Patients will be recruited into 3 successive cohorts followed by an expansion of the final cohort. For each cohort the first dose of Pembrolizumab will be given at an earlier time point during the chemo-radiation (CRT).

Pembrolizumab will be given as an IV infusion every 21 days, and a total of 8 infusions per patient at 200mg per infusion. The first dose of pembrolizumab will be given at the following times:

COHORT 1: beginning at Week 5 day 1 of CRT schedule COHORT 2: beginning at Week 3 day 1 of CRT schedule COHORT 3: beginning at Week 1 day 1 of CRT schedule** Cohort 2 will be dependent on a Safety Review Committee (SRC) recommendation. If the SRC are concerned about toxicity in Cohort 1 but not sufficiently to stop the study, they are able to recommend that Cohort 2 can change to commence pembrolizumab at week 4. If the SRC are concerned about toxicity in Cohort 2 but not sufficiently to stop the study, they are able to recommend that Cohort 3 can change to commence pembrolizumab at week 2.

Potential participants will be under the care of a consultant who specializes in the treatment of anal cancer and the patient will have been identified as requiring CRT treatment for their anal cancer. They will be assessed for eligibility before being consented and allocated to the current cohort. # Patients will be monitored for Adverse Events which will be assessed according to Common Terminology Criteria for Adverse Events (CTCAE) 4.03. Treatment guidelines are given for any immune related or infusion related events. Adverse Event review will take place weekly during CRT and at every pembrolizumab visit as well as key time during follow up.

Patient reported outcomes will be assessed using the European Organisation for Research and Treatment of Cancer (EORTC) tool during CRT, pembrolizumab treatment and follow up. Patients will be followed up for 12 months.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible for participation in this trial, the subject must:

1. Be willing and able to provide written informed consent/assent for the trial.
2. Age 18 years or over on day of signing informed consent.
3. Histologically proven Squamous Cell Cancer of Anus (SCCA) T3 / 4 N0 M0 or any N+ M0 or highly suspicious and confirmed by the MDT
4. Be willing to provide tissue sample either archival or repeat biopsy to be tested for HPV and p16.
5. Have a performance status of 0 or 1 on the ECOG Performance Scale.
6. Demonstrate adequate organ function performed within 10 days of treatment initiation:

   1. Hematological: Absolute neutrophil count (ANC) ≥1.5 x 109/L, Platelets ≥100 x 109/L,
   2. Coagulation: International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 X ULN (unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants), Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN (unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants).
   3. Renal: Serum creatinine ≤1.5 x upper limit of normal (ULN) OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≥60 mL/min for patient with creatinine levels > 1.5 x institutional ULN
   4. Hepatic Serum total bilirubin ≤ 1.5 x ULN OR Direct bilirubin ≤ ULN for patients with total bilirubin levels > 1.5 ULN
7. Female patient of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of trial medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
8. Female patients of childbearing potential must be willing to use an adequate method of contraception for the course of the trial through 120 days after the last dose of trial medication. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the patient.
9. Male patients must agree to use an adequate method of contraception starting with the first dose of trial therapy through 120 days after the last dose of trial therapy. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the patient.

Exclusion Criteria:

The subject must be excluded from participating in the trial if the subject:

1. Has malignant tumour of non-epithelial origin (sarcoma)
2. Has any metastatic disease
3. Is unsuitable for radical CRT for whatever reason
4. Is currently participating and receiving trial therapy or has participated in a trial of an investigational agent and received trial therapy or used an investigational device within 4 weeks of the first dose of treatment.
5. Has a diagnosis of immunodeficiency (see 18. For patients with HIV who may be eligible) or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
6. Has a known history of active TB (Bacillus Tuberculosis)
7. Hypersensitivity to pembrolizumab or any of its excipients.
8. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
9. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   1. Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   2. Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
10. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer or previous VIN (vulval intra-epithelial neoplasia) or vulval cancer adequately treated, or previous adequately treated breast cancer / DCIS > 5 years ago.
11. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
12. Has known history of, or any evidence of active, non-infectious pneumonitis.
13. Has an active infection requiring systemic therapy.
14. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
15. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
16. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
17. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
18. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
19. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g. HCV RNA is detected). Testing only required if patient has a history of either of these.
20. Has received a live vaccine within 30 days of planned start of study therapy. (Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability- 30 days post CRT | 30 days post chemoradiotherapy
  To assess safety of different schedules of exposure to pembrolizumab, an immune checkpoint inhibitor, concomitantly with standard CRT in patients with locally advanced T 3/4 anal cancer. Grade 3 to 5 treatment related adverse events (CTCAE - v.4.03) will be reported at 30 days post chemoradiotherapy.
Safety and tolerability- 6 weeks post CRT | 6 weeks post chemoradiotherapy
  To assess the safety of different schedules of exposure to pembrolizumab, an immune checkpoint inhibitor, concomitantly with standard CRT in patients with locally advanced T3/4 anal cancer. Grade 3 to 5 treatment related adverse events (CTCAE v.4.03) will be reported at 6 weeks post chemoradiotherapy.
Safety and tolerability - 12 weeks post CRT | 12 weeks post chemoradiotherapy
  To assess the safety of different schedules of exposure to pembrolizumab, an immune checkpoint inhibitor, concomitantly with standard CRT in patients with locally advanced T3/4 anal cancer. Grade 3 to 5 treatment related adverse events (CTCAE v.4.03) will be reported at 12 weeks post chemoradiotherapy.
Safety and tolerability - 6 months post CRT | 6 months post chemoradiotherapy
  To assess the safety of different schedules of exposure to pembrolizumab, an immune checkpoint inhibitor, concomitantly with standard CRT in patients with locally advanced T3/4 anal cancer. Grade 3 to 5 treatment related adverse events (CTCAE v.4.03) will be reported at 6 months post chemoradiotherapy.
Safety and tolerability- 9 months post CRT | 9 months post chemoradiotherapy
  To assess the safety and of different schedules of exposure to pembrolizumab, an immune checkpoint inhibitor, concomitantly with standard CRT in patients with locally advanced T3/4 anal cancer. Grade 3 to 5 treatment related adverse events (CTCAE Adverse Events v.4.03) will be reported at 9 months post chemo-radiotherapy.
Safety and tolerability- 12 months post CRT | 12 months post chemoradiotherapy
  To assess the safety of different schedules of exposure to pembrolizumab, an immune checkpoint inhibitor, concomitantly with standard CRT in patients with locally advanced T3/4 anal cancer. Grade 3 to 5 treatment related adverse events (CTCAE v.4.03) will be reported at 12 months post chemoradiotherapy.

SECONDARY OUTCOMES:
Adherence to protocol treatment | Up to 6 months post chemoradiotherapy
  Adherence to protocol treatment will be assessed by numbers of patients receiving per protocol treatment, dose delays, treatment reductions, treatment discontinuation and documenting the reasons for delays or discontinuation for each patient.
Recruitment | 2 years
  Recruitment rate will be assessed by the number of days study is open for recruitment, the number of patients screened, the number of screened patients not recruited and why and the number (proportion) of patients recruited.
Retention | Up to 12 months post chemoradiotherapy
  Retention will be assessed by the proportion of patients withdrawing from protocol treatment and number of patients lost to follow-up with documentation of reasons in each case.
Study eligibility | 2 years
  Study eligibility will be assessed by the number of patients eligible and ineligible at screening and reasons for ineligibility.
Clinical response assessment - 3 months post CRT | 3 months post chemoradiotherapy
  Clinical response assessment will be measured by RECIST v 1.1 (MRI) for the overall response rate (ORR) at 3 months post chemoradiotherapy.
Clinical response assessment - 6 months post CRT | 6 months post chemoradiotherapy
  Clinical response assessment will be measured by RECIST v 1.1 (MRI) for the overall response rate (ORR) at 6 months post chemoradiotherapy.
Clinical response assessment - 12 months follow up | 12 months follow up
  Clinical response assessment will be measured by RECIST v 1.1 (MRI) for the overall response rate (ORR) at 12 months follow up
Imaging response - 3 months post CRT | 3 months post chemo-radiotherapy
  Imaging response will be assessed by Tumor Regression Grade MRI by changes in Apparent Diffusion Coefficient (ADC) on DW sequences. Immune related modified RECIST assessments (MRI) at 3 months post chemoradiotherapy.
Imaging response - 6 months post CRT | 6 months post chemoradiotherapy
  Imaging response will be assessed by Tumor Regression Grade MRI by changes in Apparent Diffusion Coefficient (ADC) on DW sequences. Immune related modified RECIST assessments (MRI) at 6 months post chemoradiotherapy.
Imaging response - 12 months follow up | 12 months follow up
  Imaging response will be assessed by Tumor Regression Grade MRI by changes in Apparent Diffusion Coefficient (ADC) on DW sequences. Immune related modified RECIST assessments (MRI) at 12 months follow up.
Patient reported outcome - up to 6 months post CRT | Up to 6 months post chemoradiotherapy
  Patient-reported outcomes (PRO) will be measured by using the EORTC quality of life questionnaires during CRT and 6 months post-CRT.
Patient reported outcome - 12 months follow up | 12 months follow up
  Patient-reported outcomes (PRO) will be measured by using the EORTC quality of life questionnaires at 12 months follow up

CONTACTS AND LOCATIONS:
Overall Officials: Richard Adams, Prof, Principal Investigator — Velindre University NHS Trust; Mark Harrison, Dr, Principal Investigator — East and North Hertfordshire NHS Trust
Locations (11):
- Oslo University Hospital, Oslo, Norway
- United Kingdom (10):
  - Aberdeen Royal Informary, Aberdeen, Scotland
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Velindre Cancer Centre, Cardiff
  - East Suffolk and North Essex NHS Foundation Trust, Colchester
  - The Leeds Teaching Hospitals NHS Trust, Leeds
  - The Christie NHS Foundation Trust, Manchester
  - Mount Vernon Cancer Centre, Northwood
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - Swansea Bay University Local Health Board, Swansea

IPD SHARING:
Plan to Share IPD: Undecided